CLINICAL TRIAL: NCT03272789
Title: Onco-coaching of Sport-inspired for the Social, Professional and Psychological Restoring of the Patients in Cancer Remission After Allogeneic Transplantation of Hematopoietic Stem Cells: Pilot Study
Brief Title: Onco-coaching of Sport-inspired for the Social, Professional and Psychological Restoring of the Patients in Cancer Remission After Allogeneic Transplantation of Hematopoietic Stem Cells
Acronym: REBOND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REBOND-IPC 2016-014
Record Dates: First submitted 2017-08-21; First posted 2017-09-06 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Haematologic Disease (Cancer); Onco-coaching of Sport- Inspirated
MeSH Terms: conditions — Hematologic Diseases; Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interviews and questionnaires (Other): Realization of interviews (at day 0, and at 1, 2, 3 6 and 12 months) and questionnaires delivery (at day 0, and at 3, 6 and 12 months)
  Interventions: Other: Interviews with coach

INTERVENTIONS:
Other: Interviews with coach — For Interviews : done at Day 0 and at 1, 2, 3, 6 and 12 months. Questionnaires : given at Day 0, and at 3, 6 and 12 months.
  Other Names: questionnaires given by coach

SUMMARY:
Sometimes, certain patients, while the treatment comes to an end and while a remission is possible, present psychological and emotional difficulties. The return in a " new life " is lived as a factor of often unexpected stress which force the patients, from the end of the treatment, to reconsider their future orientation, their roles and social identities, their interpersonal relations, and the quality of their life.

Often, they feel a strong feeling of isolation and a shape of social marginalization stressed by the fact that forgiveness lead automatically to a spacing of the stays to the hospital, which were for them a source of social interactions. Often incapable to deal with these negative emotional situations, they live profound depressive episodes known to be associated to a lesser survival.

The investigators think that a support of type onco-coaching of sport- inspirated could allow these survivors to find a certain quality of life to see certain well-being.

In a recent study, It was analyzed the leadership " which works " in the high-level sport in France. Five selectors of national teams of team sports were questioned about their conceptions on the best practices of management and management of the people. They grant a quite particular attention on the individual consideration of the athlete and the implementation of a relationship of trust, to the delegation of the power and the sharing regulated by the decision-making which strengthen the sportsman in a feeling of autonomy and skill, catalysts of an intrinsic motivation.

These needs were satisfied, they give meaning to the share and get a psychological well-being. The satisfaction of these needs is generally made through the realization of purposes, results wished by an action, which can sometimes enter in contradiction with the satisfaction of the fundamental needs and thus damage the well-being. The role of the coach is to help the coached to target its purposes, to decide on a strategy to affect him and keep an intact motivation throughout the process. Without being therapeutic, the questioning and the action of the coach would allow the coached to reach gradually the satisfaction of its fundamental psychological needs and thus a real well-being.

The intention is to make them benefit knowledge and expertise in the field of the coaching and by a logic of research inter disciplinary to set up steps of support individualized to propose adapted answers and assist them at best in their company on returning to the life by making a significant contribution with the patients to help them to find of the autonomy in their own decision-making, to find their social identity (refusal and discharge of positive or negative discrimination), to accompany the therapeutic education of the patient towards a stake in social reeducation and finally, to highlight and to strengthen its interests and social concerns.

In terms of public health, this approach, facilitating the transition of the treatment in the complete remission, could be subjected and so improve the quality of the services of support proposed until then.

If the hypotheses of research see each other confirmed, this device coaching of sport-inspired of the patients in remission could then be transferable in other oncologic fields.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and presenting a good understanding and a practice of the French language,
* Having been treated by allogeneic transplantation of hematopoietic stem cells,
* Written informed consent,
* Affiliation to Social Security System.

Exclusion Criteria:

* Patient with a graft versus host disease requiring a treatment by immunosuppressors to be controlled,
* Patient under treatments du to complications (infections, graft versus host disease (GVHD), …),
* Patient with evolutive hematologic disease or in relapse,
* Patients deprived of liberty or placed Under the authority of a tutor,
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol or follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-07-12 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Estimate the patient's interest with this proposal of care | At inclusion
  The evaluation of this intervention will be the acceptance by the patient of the inclusion in this pilot study, and thus the percentage of the patients realizing the first appointment of onco-coaching.
  The proposal of the sessions of coaching will be made by the doctor.

SECONDARY OUTCOMES:
Estimate the improvement of the well-being of the patients at the stemming from the sessions of coaching by means of questionnaires questioning their feeling. | From inclusion to month 12
  Demonstrate an improvement of the feeling of personal efficiency with questionnaires (Generalized Self-Efficacy Scale)
Estimate the improvement of the well-being of the patients at the stemming from the sessions of coaching by means of interviews questioning their feeling. | From inclusion to month 12
  Demonstrate an improvement of the feeling of personal efficiency with interviews
Estimate the improvement of the well-being of the patients at the stemming from the sessions of coaching by means of interviews questioning their feeling. | From inclusion to month 12
  Demonstrate an improvement of the feeling of the hope with interviews
Estimate the improvement of the well-being of the patients at the stemming from the sessions of coaching by means of questionnaires questioning their feeling. | From inclusion to month 12
  Demonstrate an improvement of the feeling of the hope questionnaires (scale of the hope)
Estimate the improvement of the well-being of the patients at the stemming from the sessions of coaching by means of interviews questioning their feeling. | From inclusion to month 12
  Demonstrate an improvement of the feeling of the global motivation with interviews
Estimate the improvement of the well-being of the patients at the stemming from the sessions of coaching by means of questionnaires questioning their feeling. | From inclusion to month 12
  Demonstrate an improvement of the feeling of the global motivation with questionnaires (global motivation scale)
Estimate the improvement of the well-being of the patients at the stemming from the sessions of coaching by means of interviews questioning their feeling. | From inclusion to month 12
  Demonstrate an improvement of the quality of their interpersonal relations of the patients with interviews
Estimate the improvement of the well-being of the patients at the stemming from the sessions of coaching by means of questionnaires questioning their feeling. | From inclusion to month 12
  Demonstrate an improvement of the quality of their interpersonal relations of the patients with questionnaires (scale of the quality of the interpersonal relations)

CONTACTS AND LOCATIONS:
Overall Officials: BLAISE Didier, MD, PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- GENRE, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Institut PAOLI-CALMETTES — http://www.institutpaolicalmettes.fr